CLINICAL TRIAL: NCT07000240
Title: Pushing Using Real-time Sonographic Ultrasound Education (PURSUE)
Brief Title: Pushing Using Real-time Sonographic Ultrasound Education
Acronym: PURSUE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Anderson Gloria, Assistant Professor in Midwifery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ID 7591
Record Dates: First submitted 2025-05-20; First posted 2025-06-02 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Transperineal Ultrasound; Midwife-led Pushing Training Program; Duration of the Second Stage; Coactivation Rates of Pelvic Floor Muscles; Maternal Satisfaction; Perineal Tear Rates

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midwife-led pushing training only group (Active Comparator): The pushing training program consists of a two-hour in-person session, structured as follows:
  * 30 minutes of theoretical instruction, covering the physiological mechanisms of labor, the role of the levator ani muscle (LAM) during pushing, and optimal pushing techniques.
  * 30 minutes of practical exercises, during which women will be guided through breathing techniques, pushing strategies, and perineal relaxation.
  Interventions: Other: Midwife-led pushing training only group
- Midwife-led ultrasound-guided pushing training group (Experimental): The pushing training program consists of a two-hour in-person session, structured as follows:
  * 30 minutes of theoretical instruction, covering the physiological mechanisms of labor, the role of the levator ani muscle (LAM) during pushing, and optimal pushing techniques.
  * 30 minutes of practical exercises, during which women will be guided through breathing techniques, pushing strategies, and perineal relaxation.
  Women randomized to the ultrasound-guided pushing training group will receive additional transperineal ultrasound (TPU) evaluations during practical exercises, performed by a midwife trained in ultrasound imaging. These assessments will ensure effective LAM relaxation during pushing practices and provide real-time visual feedback to optimize muscle coordination.
  Interventions: Other: Midwife-led ultrasound-guided pushing training group

INTERVENTIONS:
Other: Midwife-led ultrasound-guided pushing training group — The pushing training program consists of a two-hour in-person session, structured as follows:
  * 30 minutes of theoretical instruction, covering the physiological mechanisms of labor, the role of the levator ani muscle (LAM) during pushing, and optimal pushing techniques.
  * 30 minutes of practical exercises, during which women will be guided through breathing techniques, pushing strategies, and perineal relaxation.
  Women randomized to the ultrasound-guided pushing training group will receive additional transperineal ultrasound (TPU) evaluations during practical exercises, performed by a midwife trained in ultrasound imaging. These assessments will ensure effective LAM relaxation during pushing practices and provide real-time visual feedback to optimize muscle coordination.
  Arms: Midwife-led ultrasound-guided pushing training group
Other: Midwife-led pushing training only group — The pushing training program consists of a two-hour in-person session, structured as follows:
  * 30 minutes of theoretical instruction, covering the physiological mechanisms of labor, the role of the levator ani muscle (LAM) during pushing, and optimal pushing techniques.
  * 30 minutes of practical exercises, during which women will be guided through breathing techniques, pushing strategies, and perineal relaxation.
  Arms: Midwife-led pushing training only group

SUMMARY:
The study aims to assess whether the use of ultrasound during a pushing lesson can facilitate easier and safer childbirth. The research will be conducted at a single hospital and will involve pregnant women in their second trimester who enroll in an online childbirth course. Participants will be randomly assigned to one of two groups:

One group will receive standard pushing instructions from a midwife.

The other group will receive the same instructions along with a brief ultrasound session to visually support correct pushing techniques.

The primary outcome is a potential reduction in the duration of the second stage of labor (when the baby is being delivered). Secondary outcomes include improved coordination of pelvic floor muscles, fewer perineal tears, a higher rate of vaginal births, reduced postnatal urinary incontinence, and greater maternal satisfaction.

Approximately 136 women will be enrolled in the study (accounting for potential dropouts). The expectation is that this integrated teaching approach will enhance the effectiveness, safety, and overall experience of pushing during labor for both mothers and their newborns.

DETAILED DESCRIPTION:
This single-center, open-label, parallel-group randomized controlled trial aims to evaluate whether integrating transperineal ultrasound into a midwife-led pushing training program can reduce pelvic floor muscle coactivation during childbirth. Pregnant women in their second trimester, recruited from an online pre-childbirth course at Fondazione Policlinico Agostino Gemelli IRCCS, will be randomized to receive either standard midwife-led training or additional ultrasound-guided instruction. The primary outcome is the reduction in the duraction of the second stage of labour, with secondary outcomes including coactivation rates of pelvic floor muscles at delivery, maternal satisfaction, perineal tear rates, vaginal delivery rates, and postpartum urinary incontinence. With an estimated sample size of 136 participants accounting for a 15% dropout, the study anticipates that ultrasound-guided training will improve pushing efficiency, decrease pelvic trauma, and enhance delivery outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women in their second trimester (approximately 14-28 weeks of gestation).
2. Willingness to participate in the preparation training program on pushing techniques.
3. Singleton pregnancy.
4. Age 18 years or older.
5. Ability to understand and provide informed consent in Italian.
6. Plan to deliver at the Fondazione Policlinico Agostino Gemelli IRCCS.

Exclusion Criteria:

1. Multifetal (e.g., twins, triplets) pregnancies.
2. Known obstetric complications or conditions that contraindicate a vaginal delivery (e.g., placenta previa).
3. Medical or psychiatric conditions that would prevent participation in the educational program or adherence to study protocols.
4. History of pelvic floor surgery or severe pelvic floor dysfunction that might affect participation or outcomes.
5. Inability to understand study requirements or provide informed consent.
6. Participants already enrolled in conflicting clinical trials or interventions that could influence the study's outcomes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Change of duration of the second stage of labor | Measured from the onset of active labor until the moment of birth.
  Change in duration (minuts) of the second stage of labor in the experimental arm compared with the control arm, defined as the elapsed time between complete cervical dilation and fetal expulsion.

SECONDARY OUTCOMES:
Levator ani muscle (LAM) coactivation rates | Measured from the onset of active labor until the moment of birth
  The levator ani muscle (LAM) coactivation rates were measured using transperineal ultrasound, evaluating the anteroposterior diameter (APD) of the levator hiatus at rest, during maximum pelvic floor muscle contraction, and during maximum Valsalva maneuver (both before and after visual feedback), with LAM coactivation defined as a reduction in APD on Valsalva compared to the resting state.
Women's satisfaction | Measured after childbirth
  Women's satisfaction with the childbirth experience and with the training program, measured through the Associazione dei Ginecologi Italiani (AGOI) women's satisfaction with childbirth care Likert Scale.
Rate of perineal tears | Baseline
  Rates of perineal tears, measured as the proportion of women experiencing perineal lacerations of any degree
Vaginal delivery rates | Baseline
  Vaginal delivery rates, measured as the proportion of women who achieved spontaneous or assisted vaginal birth (including vacuum or forceps-assisted delivery), excluding cesarean sections, as documented in the delivery records.
Operative delivery rates | Baseline
  Operative delivery rates, measured as the proportion of women who required instrumental assistance for vaginal birth, including vacuum or forceps-assisted delivery, excluding spontaneous vaginal and cesarean deliveries, as documented in the delivery records.
Urinary incontinence rates | Measured at 6 and 12 weeks postpartum
  Urinary incontinence rates at 6 and 12 weeks postpartum, measured as the proportion of women reporting involuntary leakage of urine during activities such as coughing, sneezing, or exertion (stress urinary incontinence) or experiencing a sudden, strong urge to urinate (urge incontinence), as assessed through clinical evaluation at follow-up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Ostetricia e Patologia Ostetrica, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP